CLINICAL TRIAL: NCT04135846
Title: A Focus on Alpha-1 Blockade as a Novel Pharmacological Treatment for AUD
Brief Title: Alpha-1 Blockade for Alcohol Use Disorder (AUD)
Acronym: DOXY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Carolina L Haass-Koffler, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1907002490
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol use disorder, stress
MeSH Terms: conditions — Alcoholism | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- doxazosin (Experimental): 16 mg, or maximum tolerated dose (MTD)
  Interventions: Drug: Doxazosin
- placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxazosin — 16 mg or maximum tolerated dose (MTD)
  Other Names: Cardura
  Arms: doxazosin
Drug: Placebo — Matching placebo
  Arms: placebo

SUMMARY:
The goal of this research is to replicate findings previously conducted in a pilot trial and to understand, mechanistically, the role of stress in the development of AUD pharmacotherapies that target noradrenergic blockade.

DETAILED DESCRIPTION:
16 week, between-subject, double-blind, randomized clinical trial (RCT) with doxazosin (16 mg, or maximum tolerated dose, MTD) compared to placebo in 184 treatment seeking individuals with AUD

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age
* Meet the DSM-5 criteria for AUD
* Desire to reduce or quit alcohol drinking
* Breath alcohol (BrAC) = 0.00 at each visit
* In good health as confirmed by medical history, physical examination and lab tests
* Willing to adhere to the study procedures
* Understand informed consent and questionnaires in English at an 8th grade level

Exclusion Criteria:

* Women who are breastfeeding or /positive urine test for pregnancy
* CrCl<60mL/min
* Suicide attempt in the last three months
* Current diagnosis of other substance disorder other than nicotine as assessed by self-report and urine toxicology screen at baseline
* Current use of medication that may interact with doxazosin and/or yohimbine
* History of allergy to any alpha receptor blockers
* Clinical Institute Withdrawal Assessment for Alcohol revised (CIWA-Ar) score ≥ 8
* Treatment with disulfiram, naltrexone, acamprosate, topiramate within 1 month prior to screening
* Treatment with any alpha-blocker
* Individuals with cardiac heat failure (CHF), as assessed by the medical history, the physical exam and the ECG.
* Baseline hypotension defined as BP reading lower than 90/60 mmHg
* Use of phosphodiesterase inhibitors (PDE5) erectile dysfunction medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | 6 weeks
  Number of drinks per week (DPW) in naturalistic condition as measured by the timeline follow-back (TLFB)

SECONDARY OUTCOMES:
Alcohol craving | one day
  We will measure alcohol craving using the Alcohol Craving Questionnaire (ACQ) after a cue-reactivity
Alcohol craving | six weeks
  Alcohol craving in naturalistic condition will be measured using craving the Obsessive Compulsive Drinking Scale (OCDS)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina L Haass-Koffler, PHARMD, PHD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haass-Koffler CL, Goodyear K, Zywiak WH, Magill M, Eltinge SE, Wallace PM, Long VM, Jayaram-Lindstrom N, Swift RM, Kenna GA, Leggio L. Higher pretreatment blood pressure is associated with greater alcohol drinking reduction in alcohol-dependent individuals treated with doxazosin. Drug Alcohol Depend. 2017 Aug 1;177:23-28. doi: 10.1016/j.drugalcdep.2017.03.016. Epub 2017 May 16. PMID 28551590
- [Background] Kenna GA, Haass-Koffler CL, Zywiak WH, Edwards SM, Brickley MB, Swift RM, Leggio L. Role of the alpha1 blocker doxazosin in alcoholism: a proof-of-concept randomized controlled trial. Addict Biol. 2016 Jul;21(4):904-14. doi: 10.1111/adb.12275. Epub 2015 Jun 2. PMID 26037245